CLINICAL TRIAL: NCT00255021
Title: Immunogenicity and Safety of Sanofi Pasteur Pentaxim Combined Vaccine in Infants in Thailand
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: E2I34
Record Dates: First submitted 2005-11-15; First posted 2005-11-17 (Estimated); Last update posted 2012-04-16 (Estimated); Status verified 2012-04

CONDITIONS: Diphtheria; Tetanus; Poliomyelitis; Haemophilus Infections; Pertussis
Keywords: Diphteria; Tetanus; Pertussis; Poliomyelitis; Haemophilus influenzae type b; acellular
MeSH Terms: conditions — Diphtheria; Tetanus; Poliomyelitis; Haemophilus Infections; Whooping Cough | interventions — Tetanus Toxoid; Pentavac

ARMS (1):
- 1 (Experimental)
  Interventions: Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib Vac

INTERVENTIONS:
Biological: Diphtheria, Tetanus, Polio, Acellular Pertussis and Hib Vac — 0.5 mL, IM
  Other Names: PENTAXIM

SUMMARY:
The present clinical study will assess the immunogenicity and reactogenicity of Sanofi Pasteur's DTacP-IPV// PRP~T combined vaccine (Pentavac™ or Pentaxim™) as a three-dose primary vaccination at 2, 4, and 6 months of age followed by a booster dose during the second year of life and concomitant hepatitis B vaccine at 2 and 6 months of age in infants in Thailand.

ELIGIBILITY:
Inclusion Criteria:

* Aged 53 to 70 days inclusive on the day of inclusion

Exclusion Criteria:

* Participation in another clinical trial in the 4 weeks preceding the (first) trial vaccination
* Planned participation in another clinical trial during the present trial period
* Congenital or acquired immunodeficiency; immunosuppressive therapy such as long-term systemic corticosteroid therapy.
* Systemic hypersensitivity to any of the vaccine components or history of a life threatening reaction to the trial vaccine or a vaccine containing the same substances
* Chronic illness at a stage that could interfere with trial conduct or completion.
* Blood or blood-derived products received in the past.
* Mother known as seropositive to HIV or hepatitis B
* Any vaccination in the 5 weeks preceding the first trial vaccination (except Bacille Calmette-Guerin [BCG])
* History of diphtheria, tetanus, pertussis, poliomyelitis, Haemophilus influenzae type b infection or hepatitis B (confirmed either clinically, serologically or microbiologically).
* Previous vaccination against the diphtheria, tetanus, pertussis, poliomyelitis diseases or Haemophilus influenzae type b infection with the trial vaccine or another vaccine.
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* History of/current seizures
* Febrile illness (rectal temperature ≥ 38.0°C or axillary temperature ≥ 37.4°C) or acute illness on the day of inclusion.

Ages: 2 Months to 2 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 186 (Actual)
Dates: Start 2005-12; Primary Completion 2007-09 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Immunogenicity: To provide information concerning the immune response of the DTacP-IPV//PRP~T combined vaccine | 1 month post-vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Sanofi Pasteur, a Sanofi Company
Locations (1):
- Bangkok, Thailand

REFERENCES:
- See also: Related Info — http://www.sanofipasteur.com